CLINICAL TRIAL: NCT06685952
Title: The Application of Ultrasonic Measurement of Optic Nerve Sheath Diameter in Liposuction Surgery
Status: Completed | Type: Observational
Sponsor: The Plastic Surgery Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College (Other)
Responsible Party: Principal Investigator, Xu Wenli, Attending physician, The Plastic Surgery Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College
Other Study IDs: ZX2024310
Record Dates: First submitted 2024-11-07; First posted 2024-11-13 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Optic Nerve Sheath Diameter
Keywords: Optic nerve sheath diameter; Sedation and analgesia anesthesia; Liposuction surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prone position group: Sedation and analgesia anesthesia will be administered after the prone position.
  All patients will receive standardized sedation and analgesia anesthesia with 1ug/kg sufentanil，1ug/kg/h dexmedetomidine，1mg/h midazolam，0.05-0.1ug/kg/min remifentanil. And adjust the drug speed according to the patient's respiratory rate, BIS changes.
  Optic nerve sheath diameter (ONSD), carotid artery flow rate, Bispectral index (BIS), liposuction swelling fluid input, infusion volume, end-expiratory carbon dioxide, mean arterial pressure, heart rate, peripheral oxygen saturation, body temperature and respiratory rate will be measured at four time points respectively.
- Supine group: Sedation and analgesia anesthesia will be administered after the supine position.
  All patients will receive standardized sedation and analgesia anesthesia with 1ug/kg sufentanil，1ug/kg/h dexmedetomidine，1mg/h midazolam，0.05-0.1ug/kg/min remifentanil. And adjust the drug speed according to the patient's respiratory rate, BIS changes.
  Optic nerve sheath diameter (ONSD), carotid artery flow rate, Bispectral index (BIS), liposuction swelling fluid input, infusion volume, end-expiratory carbon dioxide, mean arterial pressure, heart rate, peripheral oxygen saturation, body temperature and respiratory rate will be measured at four time points respectively.

SUMMARY:
The main purpose of this study is to investigate the effect of changes in Optic Nerve Sheath Diameter (ONSD) measured at different operating position during Liposuction Surgery.

Optic nerve sheath diameter (ONSD) has been shown to be a noninvasive indicator for monitoring intracranial pressure changes.

The use of anesthetic drugs will reduce the intracranial pressure. However, prone position and large fluid infusion can still lead to increased intracranial pressure.

The investigators hypothesized that during sedation and analgesia anesthesia, patients in prone position had higher ONSD.

DETAILED DESCRIPTION:
Liposuction is a common type of surgery in plastic surgery. In this type of surgery, the position is often changed from prone to supine. Different surgical positions, especially excessive flexion or rotation of the neck, can cause compression of the internal jugular vein, resulting in blocked cerebral venous return and resulting in increased intracranial pressure. Sedation and analgesia anesthesia are often used in liposuction surgery to provide the patient with an appropriate depth of anesthesia, preserve the patient's independent breathing, and can wake the patient during the operation to complete the position switch independently. Dexmedetomidine is a commonly used drug for sedation and analgesia anesthesia. Studies have reported that dexmedetomidine can be used to control intracranial pressure in special surgical positions by reducing cerebral metabolic rate, maintaining cerebral oxygen supply and demand balance, shrinking cerebral vessels and other functions.

Other studies have suggested that IOP increases during prone anesthesia, despite the effect of anesthetic drugs on lowering IOP. IOP, choroidal thickness, and optic nerve diameter also increased in normally awake patients in prone position. Optic nerve sheath diameter (ONSD) has been shown to be a noninvasive indicator of intracranial pressure changes and an independent factor of mortality, poor prognosis, and severity of traumatic brain injury. ONSD measurement is often used in laparoscopic surgery under general anesthesia to observe the effect of elevated CO2 in pneumoperitoneum on IOP. The changes of intracranial pressure were evaluated by ONSD when the head was low and the feet were high.

At present, there are no studies to observe the change of ONSD at different positions during Liposuction Surgery with sedation and analgesia.

The investigators hypothesized that during sedation and analgesia anesthesia, patients in prone position had higher ONSD.

This is an observational study. They were divided into two groups according to the operation, prone group and supine group.T0 awake, T1 30min after sedation and analgesia, T2 30 minutes after T1， T3 end of the operation. Record Optic nerve sheath diameter (ONSD), carotid artery flow rate, Bispectral index (BIS), liposuction swelling fluid input, infusion volume, end-expiratory carbon dioxide, mean arterial pressure, heart rate, peripheral oxygen saturation, body temperature and respiratory rate. Statistically significant differences were assessed.

The incidence of headache, nausea, vomiting and delirium were observed within 24 hours after operation.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-50 years, undergoing liposuction surgery.
* American Society of Anesthesiologists (ASA) physical status Ⅰ and Ⅱ.
* Voluntary participation and signed an informed consent form.

Exclusion Criteria:

* Uncontrolled hypertension, diabetes.
* High nearsightedness or farsightedness, recent eye surgery, and other conditions in which ONSD cannot be measured.
* Moderate to severe obstructive sleep apnea syndrome was present before surgery.
* History of severe mental or neurological diseases, drug or psychotropic drug abuse.
* Cognitive dysfunction or inability to communicate.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Female patients who will undergo liposuction surgery under sedation and sedative anesthesia. Fat suction areas can be the abdomen, lower back, limbs and other parts.
Sampling Method: Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2024-11-19 (Actual); Primary Completion 2025-05-25 (Actual); Study Completion 2025-05-26 (Actual)

PRIMARY OUTCOMES:
Optic nerve sheath diameter | Enter the operating room, 30min and 60min after sedative AND analgesic anaesthesia, end of surgery
  Optic nerve sheath diameter under Ultrasonic measurement

SECONDARY OUTCOMES:
Carotid artery flow rate | Enter the operating room, 30min and 60min after sedative AND analgesic anaesthesia, end of surgery
  Peak systolic velocity (PSV), End-diastolic blood flow velocity (EDV) under Ultrasonic measurement
Carotid artery width | Enter the operating room, 30min and 60min after sedative AND analgesic anaesthesia, end of surgery
  Carotid artery flow rate under Ultrasonic measurement
Bispectral index (BIS) | 30min and 60min after sedative AND analgesic anaesthesia, end of surgery
  Anesthesia depth measurement. 50-70 means appropriate level of sedation
OAA/S score | 30min and 60min after sedative AND analgesic anaesthesia, end of surgery
  Observer's assessment alert/Sedation. 1-5, 2-3 means a better outcome
Liposuction swelling fluid input | 30min and 60min after sedative AND analgesic anaesthesia, end of surgery
  Amount of swelling anesthetic injected into fat suction area
Infusion volume | 30min and 60min after sedative AND analgesic anaesthesia, end of surgery
  Intraoperative intravenous fluid infusion
Urine volume | 30min and 60min after sedative AND analgesic anaesthesia, end of surgery
  Intraoperative urine drainage
Systolic blood pressure (SBP) | Enter the operating room, 30min and 60min after sedative AND analgesic anaesthesia, end of surgery
  Intraoperative hemodynamics
Diastolic blood pressure (DBP) | Enter the operating room, 30min and 60min after sedative AND analgesic anaesthesia, end of surgery
  Intraoperative hemodynamics
Mean blood pressure (MBP) | Enter the operating room, 30min and 60min after sedative AND analgesic anaesthesia, end of surgery
  Intraoperative hemodynamics
Heart rate (HR) | Enter the operating room, 30min and 60min after sedative AND analgesic anaesthesia, end of surgery
  Intraoperative hemodynamics
Saturation of Peripheral Oxygen (SPO2) | Enter the operating room, 30min and 60min after sedative AND analgesic anaesthesia, end of surgery
  Intraoperative vital signs
body temperature (T) | Enter the operating room, 30min and 60min after sedative AND analgesic anaesthesia, end of surgery
  Intraoperative vital signs
The partial pressure of end-tidal carbon dioxide (PetCO2) | Enter the operating room, 30min and 60min after sedative AND analgesic anaesthesia, end of surgery
  Respiratory monitoring during surgery
respiratory rate (RR) | Enter the operating room, 30min and 60min after sedative AND analgesic anaesthesia, end of surgery
  Respiratory monitoring during surgery
Postoperative adverse events | Day 1 after surgery
  Number of Participants with postoperativ headache, nausea AND vomiting (PONV)

CONTACTS AND LOCATIONS:
Overall Officials: Dong Yang, Study Chair — Plastic Surgery Hospital, Chinese Academy of Medical Sciences and PekingUnion Medical College
Locations (1):
- Xu Wenli, Beijing, Beijing Municipality, China